CLINICAL TRIAL: NCT05515094
Title: Strengthening Women's Agency in Pregnancy (SWAP): Empowerment Counselling Intervention [ECI] for Pregnant Women and Girls Affected by Intimate Partner Violence in a Refugee Camp in Tanzania
Brief Title: Strengthening Women's Agency During Pregnancy
Acronym: SWAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Rescue Committee (Other)
Collaborators: World Health Organization (Other); George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DF222
Record Dates: First submitted 2022-05-15; First posted 2022-08-25 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-08

CONDITIONS: Intimate Partner Violence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Empowerment Counseling Intervention) (Experimental): The Empowerment Counseling Intervention (ECI) entails directly linking women to on-site case managers who will provide first-line support (i.e., a brief psychosocial support session) and a safety and health assessment to women who are attending to receive ANC and disclose violence. The intervention (e.g., the initial counselling session), adapted from current case management guidelines and the Safe and Sound intervention at health facilities, will be administered directly at the health facility after a woman screens positive for IPV. In line with a survivor centered approach, as part of the initial session, the survivor participant will be invited back for further counselling sessions as part of the intervention curriculum, in addition to being supported to access other services based on her preferences, such as group psychosocial support. The intervention manual acts as a guide and support for trained social workers to support the unique needs of each survivor.
  Interventions: Behavioral: Empowerment Counseling Intervention
- Standard of Care (No Intervention): Women in the comparison arm will receive the standard of care and be referred to support services at the nearby IRC Women's Protection and Empowerment (WPE) office.

INTERVENTIONS:
Behavioral: Empowerment Counseling Intervention — The intervention entails case managers conducting first-line support (i.e., a brief psychosocial support session), and a safety and health assessment, adapted from current case management content and the Safe and Sound intervention.
  Arms: Intervention Arm (Empowerment Counseling Intervention)

SUMMARY:
This research aims to address the feasibility and acceptability of a brief empowerment counselling intervention (ECI) among pregnant women and girls receiving antenatal care (ANC) who have experienced intimate partner violence (IPV), in humanitarian healthcare settings.

DETAILED DESCRIPTION:
This research aims to address the feasibility and acceptability of a brief empowerment counseling intervention (ECI) among pregnant women and girls receiving antenatal care (ANC) who have experienced intimate partner violence (IPV), in humanitarian healthcare settings. This 3- year study will take place in two IRC-managed health posts in a refugee camp in Kigoma, Tanzania. The objectives of the study are to: 1) Adapt, as needed, for use in the context of ANC in a humanitarian setting, a brief ECI to address women's and girls' exposure to sexual and/or physical IPV during pregnancy, by improving their mental health, self-efficacy, safety, and coping strategies; 2) Test the ECI through a pilot randomized controlled trial, determining whether the intervention is feasible/acceptable and whether it improves women's self-efficacy, reduces mental distress and increases uptake of longer-term IPV services; 3) Test the feasibility of integrating such an intervention into pre-existing ANC service delivery in humanitarian settings and make recommendations for future intervention research and development, including effectively linking routine enquiry of IPV in ANC settings with support service use.

ELIGIBILITY:
Inclusion Criteria:

* Women or girl aged 15 years or older:
* Pregnant (any trimester);
* Attending their 2nd or later ANC visit;
* Have experienced physical and/or sexual and/or severe psychological IPV in the past 12 months;
* Consent to participate.

Exclusion Criteria:

* At their first ANC visit or accompanied by their partner (or anyone else) at the ANC visit;
* Under age 15;
* Unable to provide informed consent/assent;
* Suicidal or at risk of severe violence or of being murdered; and/or
* In a high-risk situation or medically high risk.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire - 9 | 3 months endline survey, past two week recall period
  Depressive symptoms will be assessed via the PHQ-9 questionnaire. The range of scores is 0-27. A higher score indicates more symptoms.
General Self-Efficacy Scale | 3 months endline survey, present recall period
  Adapted measure of the GSE Scale. Possible score 10-40; higher indicating more self-efficacy.

SECONDARY OUTCOMES:
Checklist of Safety Behaviors | Through study completion, average length three months;
  12 item index of safety behaviors; increased number of safety behaviors indicates improvement in safety behaviors
Uptake of case management services | Through study completion, average length three months;
  Two items indicating whether a survivor has shared information about violence with others or has sought additional services. Higher endorsement is better uptake of case management services.
Intimate Partner violence- | Through study completion, average length three months;
  Proportion of women indicating they have experienced physical, sexual, and / or psychological IPV using the WHO multi-country study instruments on IPV

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Garcia Moreno, Principal Investigator — World Health Organization; Mary Ellsberg, Principal Investigator — George Washington University; Bathsheba Mahenge, Principal Investigator — International Rescue Committee

IPD SHARING:
Plan to Share IPD: Undecided